CLINICAL TRIAL: NCT03521297
Title: Safety and Efficacy of Probiotics in Primary Biliary Cholangitis (PBC) Patients With Poor Ursodeoxycholic Acid (UDCA) Response
Brief Title: Probiotics in PBC Patients of Poor Response to UDCA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Lin Bingliang, professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PBC-UDCA
Record Dates: First submitted 2018-04-28; First posted 2018-05-11 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Primary Biliary Cholangitis (PBC)
Keywords: Probiotics; ursodeoxycholic acid (UDCA)
MeSH Terms: conditions — Liver Cirrhosis, Biliary | interventions — Probiotics

STUDY DESIGN:
Who Masked: Investigator
Masking Description: single(Investigator)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo group (Placebo Comparator): Placebo (three times per day, one pack each time) and UDCA (13-15mg/kg/day), orally, 6 months
  Interventions: Dietary Supplement: Placebo
- Probiotics group (Experimental): Probiotics (three times per day, one pack each time) and UDCA(13-15mg/kg/day), orally, 6 months
  Interventions: Drug: Probiotic

INTERVENTIONS:
Drug: Probiotic — UDCA combined probiotic
  Other Names: Probiotic group
  Arms: Probiotics group
Dietary Supplement: Placebo — UDCA combined placebo
  Arms: Placebo group

SUMMARY:
The safety and efficacy of probiotics in primary biliary cholangitis (PBC) patients with poor ursodeoxycholic acid (UDCA) response.

DETAILED DESCRIPTION:
PBC patients with poor ursodeoxycholic acid (UDCA) response are selected and randomly assigned into probiotic group and control group. Patients in probiotic group receive probiotic(Micro V Probiotics) combined UDCA for 6 months and then continue to take UDCA alone. Patients in control group continue to take UDCA alone. Biochemical indicators, immunological indicators, liver stiffness, and ultrasound of the two groups of patients were collected. GLOBE and UK-PBC scoring system are used to assesse prognosis.The feces and serum of all patients are collected to observe the differences in fecal microbial polymorphisms in the two groups of patients. Metabolomics are used to study the differences in the bile acids and short chain fatty acid metabolites of the serum and feces of the two groups of PBC patients.

ELIGIBILITY:
Inclusion Criteria:

1. PBC patients (diagnosed with PBC according to 2009 AASLD PBC PRACTICE GUIDANCE), take UDCA more than 12 months and have poor response;
2. Age 18-70 years.

Exclusion Criteria:

1. Any other liver disesases (viral hepatitis, HIV positive, alcohol abuse, hemochromatosis, hepatolenticular degeneration, α1-antitrypsin deficiency and so on);
2. Important organ dysfunction such as heart, lung and kidney which affect the life expectancy;
3. Have congenital galactosemia, glucose malabsorption syndrome or lactase deficiency.
4. Patients allergic to research drugs or excipients;
5. Pregnant or lactating women;
6. Not signed informed consent;
7. Have antibiotics one month before enrollment;
8. Microecological preparations (probiotics, prebiotics, synbiotics, etc.) were used before the enrollment;
9. Malignant tumors, nerves and mental disorders;
10. Those who participated in other drug clinical trials in the past 3 months.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-01-20 (Estimated); Primary Completion 2021-01-31 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
Biochemical response | 6 month
  Percentage of patients with biochemical response (serum ALP(U/L) or GGT(U/L) decreased by 20% from baseline)

CONTACTS AND LOCATIONS:
Overall Officials: Bingliang Lin, MD, Study Director — Third Affliated Hospital of Sun Yat-sen University
Locations (1):
- Third Affliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No